CLINICAL TRIAL: NCT06862102
Title: Prospective Clinical Study on the Role of Multiple Human Papillomavirus Infections in Lower Genital Tract Dysplasias and Its Interactions with HPV Vaccination
Brief Title: Multiple Human Papillomavirus Infections in the Development of CIN
Acronym: HPV dysplasia
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Barbara Gardella, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: HPV-dysplasia
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: CIN - Cervical Intraepithelial Neoplasia; HPV; HPV Vaccines
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervical stripping
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CIN1 with multiple HPV genotypes infection underwent vaccination
  Interventions: Biological: HPV vaccine
- CIN1+ with multiple HPV genotypes infection not underwent vaccination

INTERVENTIONS:
Biological: HPV vaccine — vaccine administration
  Groups: CIN1 with multiple HPV genotypes infection underwent vaccination

SUMMARY:
Multiple infections of high-risk genotypes of Human Papillomavirus (HR-HPV) in patients with abnormal cervical cytological or histological findings are detectable in a percentage ranging from 20% to 50% of cases.

Some studies have detected a certain tendency to specific clustering in multiple infections, both inter-species and inter-genotypic, such as HPV 31-35-56, HPV 16-51-52, HPV 16-18, HPV 51-52. Furthermore, a greater tendency of the HPV16 genotype to cluster with genotypes of different species is reported in the literature. However, other studies claim a random character of such genotypic associations in multiple infections. This heterogeneity of results of the studies present in the literature underlies multiple factors, both epidemiological and methodological, implicated in the high variability of prevalence and diagnostic findings of multiple infections. In particular, with regard to epidemiological characteristics, factors influencing the distribution of multiple infections appear to be the origin and type of population, economic-social status, young age, HIV seropositivity and recent sexual activity. A further hypothesized element is represented by a possible individual susceptibility dictated by the immune profile of the host towards specific genotypes, potentially facilitating the occurrence of co-infections by these, possibly resulting in a synergistic effect on the oncogenic potential. From a clinical point of view, to date multiple cross-sectional studies suggest an association between multiple infections of HR-HPVs and an increased risk of high-grade cervical dysplasia. In particular, a proportional relationship is observed between the number of genotypes present and the severity of the lesion. Furthermore, it has been reported that the correlation between multiple HR-HPV infections and severe cervical dysplasia CIN2+ is significant both in the presence and absence of the known oncogenic genotype HPV16, assuming a possible synergistic interaction between specific high-risk genotypes. However, other studies seem to refute the clinical relevance of multiple infections in the risk of neoplastic progression of cervical lesions, mostly claiming the precept of "one virus, one lesion", such that each dysplastic lesion is associated with the action of a distinct HR-HPV genotype. In this assumption, therefore, it is argued that moderate-severe cervical dysplasias are due to the action of a single oncogenic genotype, predominantly HPV16, while the presence of other HR-HPVs is attributable to transient infections, mostly represented by mild dysplasias (CIN1). As far as biological knowledge is concerned, in vitro studies currently demonstrate how it is possible for a single cell to be co-infected by at least two HR-HPV genotypes and how this can result in peculiar inter-genotypic molecular interactions that influence the replication cycle and the respective capacity for cellular persistence and transformation of the individual genotypes involved. The inter-genotypic competition mechanisms detected, therefore, occur mostly during the initial phases of acute infection by the HR-HPVs involved. However, it has been demonstrated that when a persistent infection of a genotype has already been established, this is no longer able to negatively interact with a subsequent incident infection by a different HR-HPV genotype. This finding in the biological field is consistent with the clinical correlate according to which the association between multiple HR-HPV infections and the risk of high-grade cervical dysplasia is greater when these are established on a pre-existing persistent infection. Therefore, it is conceivable that there is a higher rate of genotype-specific association in multiple HR-HPV infections found in cervical dysplastic lesions, defined by the peculiar capacities of the individual genotypes to give rise to persistent cellular infections. Despite the proven efficacy of vaccination programs in preventing cervical dysplastic lesions and infection by the main viral genotypes with high oncogenic risk, numerous studies demonstrate the clinical efficacy of HPV vaccination also in reducing the rate of disease recurrence in patients undergoing excisional treatment. A first explanatory hypothesis of this phenomenon is represented by the protection that the vaccination procedure would provide to those patients not previously infected by the target HR-HPV genotypes, potentially causative of de novo infections with high oncogenic risk. A further hypothesis under study is represented by the fact that the administration of the HPV vaccine following excisional treatment would prevent the reduction of the immune response against HPV.

ELIGIBILITY:
Inclusion Criteria:

* Pap smear cytology suggestive of dysplastic cervical lesion worthy of colposcopic evaluation and HPV test
* HPV-related vaginal and/or vulvar lesion
* patients with histological diagnosis after biopsy of Cervical Intraepithelial Neoplasia (CIN) or invasive cervical cancer of stage lower than FIGO staging 1B.

Exclusion Criteria:

* pregnancy
* age less than 18 years
* previous treatment for HPV-related vaginal, vulvar or cervical lesion in the previous 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HPV infection and abnormal citology attending colposcopy
Sampling Method: Non-Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
effect of HPV vaccination on multiple HPV infection | 2 years
  To evaluate the effect of multiple HPV infections on the risk of regression, persistence or progression to CIN2/3 after 24 months from biopsy for CIN1+ in relation to the execution of HPV vaccine.

SECONDARY OUTCOMES:
progression to CIN2+ in vaccinated group | 2 years
  To compare the progression of cervical dysplasia in the population vaccinated with the anti-HPV vaccine 9 within the unvaccinated population at 2 years after excisional treatment for CIN2+ Progression is given by persistence (within 6 months) or recurrence (12 months or more).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SC Ostetricia e Ginecologia 1, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: Yes
at the end of the study
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Ghelardi A, Parazzini F, Martella F, Pieralli A, Bay P, Tonetti A, Svelato A, Bertacca G, Lombardi S, Joura EA. SPERANZA project: HPV vaccination after treatment for CIN2. Gynecol Oncol. 2018 Nov;151(2):229-234. doi: 10.1016/j.ygyno.2018.08.033. Epub 2018 Sep 6. No abstract available. PMID 30197061
- [Background] Spinillo A, Gardella B, Roccio M, Alberizzi P, Cesari S, Patrizia M, Silini E. Multiple human papillomavirus infection with or without type 16 and risk of cervical intraepithelial neoplasia among women with cervical cytological abnormalities. Cancer Causes Control. 2014 Dec;25(12):1669-76. doi: 10.1007/s10552-014-0471-6. Epub 2014 Oct 9. PMID 25296710